CLINICAL TRIAL: NCT05619731
Title: Deployment of Teleconsulting in Geriatric Oncology for Patients Aged 75years or Older Initiating an Oncologic Treatment and Living in Remote Area With no or Few Access to Geriatric Oncology Evaluation Nearby Their Oncologic Treatment Center
Brief Title: Deployment of Teleconsulting in Geriatric Oncology for Older Patients
Acronym: TeleOncoGe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RCAPHM21_0428; 2021-A02984-37 (Registry Identifier: IdRCB)
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: Older adults; Telemedecine; Cancer; Pharmaceutical expertise; Comprehensive Geriatric Assessment; Unexplained re-hospitalization
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm with oncology tele-consultation and pharmaceutical tele-expertise (Experimental): patients will benefit from geriatric oncology tele-consultation and pharmaceutical tele-expertise
  Interventions: Other: Geriatric oncology tele-consultation and pharmaceutical tele-expertise
- Conventional care (No Intervention): patients will benefit from conventional care

INTERVENTIONS:
Other: Geriatric oncology tele-consultation and pharmaceutical tele-expertise — tele consultation
  Arms: Experimental arm with oncology tele-consultation and pharmaceutical tele-expertise

SUMMARY:
Cancer affects mostly older adults. The development of Geriatric Oncology has greatly improved the management of older patients with the Comprehensive Geriatric Assessments (CGA) being conducted before cancer treatment. A CGA encompasses several dimensions such as comorbidities, but also functional, nutritional or cognitive domains. The International guidelines recommended establishing cooperation with pharmacists as part of the CGA in order to review prescriptions of older patients with cancer and to avoid adverse side effects of treatment. However, the CGA before starting oncological treatment offer is limited in France, especially in some regions which are less populated, or where access to medical centers are difficult. The main objective of our work is to evaluate the impact of telemedicine in geriatric oncology consultation of unexplained re-hospitalization rate at 3 months in the acute care unit. The secondary objectives are to evaluate the impact of telemedicine on unexplained re-hospitalization rate at 6 months, on the secondary toxicities, on the postoperative complications in patients treated surgically, on the overall survival and on the acceptance of the pharmaceutical recommendations by the physicians, but also the impact of telemedicine in medico-economic terms and the satisfaction of patients and oncologists benefiting from teleconsultation.

It is a multicenter, prospective, randomized study involving 500 patients in 9 participating centers, including 6 peripheral hospitals. The experiment will be represented by the implementation of telemedicine in oncology centers where this expertise is not very available, allowing them to benefit from geriatric oncology teleconsultation and pharmaceutical tele-expertise carried out by three university hospitals. Patients recruited by oncologists, according to the inclusion criteria, will give their written consent to participate. Centers were randomized. In the control arm, patients will be treated according to the usual oncological management as defined for each type of cancer. In the interventional arm, patients will benefit from a CGA with a geriatric oncology teleconsultation as well as a pharmaceutical tele-expertise before the initiation of oncological treatment.

DETAILED DESCRIPTION:
Cancer affects nearly 50% of people over 65 years. The development of Geriatric Oncology has greatly improved the management of older patients with the Comprehensive Geriatric Assessments (CGA) being conducted before cancer treatment. A CGA encompasses several dimensions such as comorbidities, functional, nutritional or cognitive domains. This practice aims to guarantee adapted oncological treatment to their frailties through a multidisciplinary and multi-professional approach. The International guidelines recommended establishing cooperation with pharmacists as part of the CGA in order to review prescriptions of older patients with cancer and avoid adverse side effects of treatment. However, the CGA before starting oncological treatment offer is limited in France, especially in some regions which are less populated, or where access to medical centers are difficult for older patients. Telemedicine is developing in France and is particularly intended for rural populations in order to facilitate access to specialized consultations. The ongoing COVID-19 pandemic episode has clearly enabled to develop telemedicine in hospitals. The main objective of our work is to evaluate the impact of telemedicine in geriatric oncology consultation on the unexplained re-hospitalization rate at 3 months in the acute care unit. The secondary objectives are to evaluate the impact of telemedicine on the unexplained re-hospitalization rate at 6 months, on the secondary toxicities of oncological treatments, on the postoperative complications in patients treated surgically, on the overall survival and on the acceptance of the pharmaceutical recommendations by the physicians, but also on medico-economic terms and on satisfaction of patients and oncologists benefiting from teleconsultation.

It is a multicenter, prospective, randomized study involving 500 patients in 9 participating centers, including 6 peripheral hospitals. The experiment will be represented by the implementation of telemedicine in oncology centers where this expertise is not very available, allowing them to benefit from geriatric oncology teleconsultation and pharmaceutical tele-expertise carried out by three university hospitals. Patients recruited by oncologists, according to the inclusion and non-inclusion criteria, will give their written consent to participate. Centers will be randomized into two arms. In the control arm, patients will be treated according to the usual oncological management as defined for each type of cancer. In the interventional arm, patients will benefit from a CGA with a geriatric oncology teleconsultation as well as a pharmaceutical tele-expertise before the initiation of oncological treatment.

The methodology and analysis plan will be based on the criteria developed by the Consolidated Standards of Reporting Trials Statement (CONSORT) group and more specifically on the extension concerning cluster studies. The expected benefits are a reduction of unexplained re-hospitalizations rate and of inequalities concerning access to care for older patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 75 years and older
* Suffering from all types and all stages of cancer and treated for cancer in participating centers
* G8 (screening tool) ≤ 14/17
* Agreeing to benefit from a geriatric oncology assessment
* Having signed a consent
* Affiliated to French social security or a similar French solidarity scheme

Exclusion Criteria:

* Patients under guardianship or curatorship or inability to sign consent
* Patients with severe cognitive impairment (MMSE < 10/30)
* Patients with severe hearing or visual impairments as these patients will have difficulty performing the telemedicine consultation
* Patients with a significant language barrier without an interpreter present because these patients will have difficulty carrying out the Telemedicine consultation
* Patients with expectancy less than 3 months

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2027-05-18 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of telemedicine in geriatric oncology on the unexplained re-hospitalization rate at 3 months in the medicine-surgery-oncology-acute care units (with or without going through the emergency department). | Three months after inclusion
  Unexplained re-hospitalization rate at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure COUDERC, Principal Investigator — Assistance Publique des Hôpitaux de Marseille (AP-HM)
Locations (1):
- CH Avignon, Avignon, France

IPD SHARING:
Plan to Share IPD: No